CLINICAL TRIAL: NCT04874090
Title: Investigation of the Effectiveness of Dry Needle Treatment Applied to Acupuncture Points in Parkinson's Disease on Pain
Brief Title: The Effectiveness of Acupuncture Therapy on Pain in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Elif yaksi, Medical Doctor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-EY-04
Record Dates: First submitted 2021-04-12; First posted 2021-05-05 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease; Pain, Neck
MeSH Terms: conditions — Parkinson Disease; Neck Pain | interventions — Acupuncture Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: We have two groups. First group will recieve acupuncture treatment and exercise group, second group will recieve only exercise treatment
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Investigator will apply the acupuncture treatment to the first group to the neck area. BL-15, BL-18, BL-23, BL-25, KB-4, Du-20, GB-20, CV-14, KB-10, Ex-26, Yin Tang, Ah-shi points will be used. 0.25x25 mm, sterile, steel, disposable, acupuncture needle will be used for acupuncture points and painful trigger points. The treatment will be applied twice a week, on average 10 sessions. Dry needling treatment will be applied to the patients by a certified physician. All patient will be performed the neck exercises program.
  Interventions: Other: Acupuncture; Other: Exercises
- Exercises group (Other): Patients will perform only neck exercises.
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Acupuncture — Investigator will apply the acupuncture treatment to the first group to the neck area. BL-15, BL-18, BL-23, BL-25, KB-4, Du-20, GB-20, CV-14, KB-10, Ex-26, Yin Tang, Ah-shi points will be used. 0.25x25 mm, sterile, steel, disposable, acupuncture needle will be used for acupuncture points and painful trigger points. The treatment will be applied twice a week, on average 10 sessions. Dry needling treatment will be applied to the patients by a certified physician. All patient will be performed the neck exercises program
  Arms: Interventional group
Other: Exercises — Patient will perform neck exercises

SUMMARY:
Parkinson's Disease (PD) is a chronic, progressive, degenerative movement disorder that is characterized by motor and nonmotor symptoms and its incidence increases with age. It has been reported that 40-90% of patients have pain symptoms in PD. Pain can be the result of motor fluctuations, dystonic muscle contractions, deep visceral pain, and musculoskeletal pain.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a chronic, progressive, degenerative movement disorder that is characterized by motor and nonmotor symptoms and its incidence increases with age. It is the second most common neurodegenerative disease after Alzheimer's.Bradykinesia, which is characterized by rigidity, resting tremor, postural instability, gait disturbance and progressive decrease in the speed and amplitude of repetitive movements throughout the course of the disease, are the main cardinal motor findings.Sensory dysfunction such as non-motor findings in PD, disruption in the sleep-wake cycle, neuropsychiatric findings such as dementia, confusion, hallucinations, delirium, depression, gastrointestinal dysfunction, autonomic nervous system disorders such as bladder dysfunction, orthostatic hypotension, and pain perception may develop.Although dopaminergic therapies in PD are the gold standard in the treatment of disorders such as bradykinesia, rigidity and tremor, adequate response cannot be obtained in the treatment of non-motor symptoms. For this reason, rehabilitative applications, especially pain symptom, and complementary medicine methods are very important.It has been reported that 40-90% of patients have pain symptoms in PD. Pain can be the result of motor fluctuations, dystonic muscle contractions, deep visceral pain, and musculoskeletal pain.

Acupuncture and dry needling therapy have been used clinically for a long time as pain relievers such as migraine pain, low back pain, chronic pain and cancer pain. On the other hand, there are very limited and very limited number of studies on the efficacy of dry needle therapy applied to acupuncture points in pain control in PD.In this study, our aim is to investigate the effectiveness of dry needling treatment applied to acupuncture points in neck pain due to PH on musculoskeletal pains.

ELIGIBILITY:
Inclusion Criteria:

* Being Parkinson's Disease
* Age 45-75
* Have a pain due to Parkinson's Disease

Exclusion Criteria:

* Presence of advanced dementia or mental disability
* Pain due to ınflammatory conditions
* Using anticoagulant therapy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Visuel Analog Scale | Baseline
  This scale consists of a 100 mm horizontal line and is marked from 0 to 10. In our study, patients were told that the "0" point was not pain at all, and the "10" point showed unbearable pain, and patients were asked to mark their pain intensity by considering their pain at rest.
Visuel Analog Scale | 6 weeks
  This scale consists of a 100 mm horizontal line and is marked from 0 to 10. In our study, patients were told that the "0" point was not pain at all, and the "10" point showed unbearable pain, and patients were asked to mark their pain intensity by considering their pain at rest.
Neck Disability Index | Baseline
  This index consists of 10 questions and is used to evaluate how and to what extent the neck pain affects the daily life activities of the patient. Neck disability index includes the severity of pain, self-care, load-lifting, reading, headache, concentration, driving, sleep, and social activity parameters. The patients are asked to mark the most appropriate for them from the 6 options given for each parameter. Each title is scored from 0 "(no disability) to 5" (complete disability). The total score is between 0 (no disability) and 50 (total disability). After the total score is obtained, the value calculated according to the formulation is concluded as % insufficiency. High scores indicate high disability, and low scores indicate a low disability level.
Neck Disability Index | 6 weeks
  This index consists of 10 questions and is used to evaluate how and to what extent the neck pain affects the daily life activities of the patient. Neck disability index includes the severity of pain, self-care, load-lifting, reading, headache, concentration, driving, sleep, and social activity parameters. The patients are asked to mark the most appropriate for them from the 6 options given for each parameter. Each title is scored from 0 "(no disability) to 5" (complete disability). The total score is between 0 (no disability) and 50 (total disability). After the total score is obtained, the value calculated according to the formulation is concluded as % insufficiency. High scores indicate high disability, and low scores indicate a low disability level.

SECONDARY OUTCOMES:
Health Assesment Quality | Baseline
  This questionnaire consists of eight questions designed to assess the effects of individuals' health status on daily living. Day-to-day activities such as dressing, hygiene, eating, and walking are assessed, and high scores indicate poor health status.
Health Assesment Quality | 6 weeks
  This questionnaire consists of eight questions designed to assess the effects of individuals' health status on daily living. Day-to-day activities such as dressing, hygiene, eating, and walking are assessed, and high scores indicate poor health status.
MDS-Unified Parkinson's Disease Rating Scale | Baseline
  This is an extensive scale employed for the clinical evaluation of severity of PD. It consists of four sections including non-motor findings, motor problems, motor findings, and treatment complications. Fourteen motor findings (0 - no finding, or normal, 4- severe finding) in the second section of the scale and comprising the motor problems part.
MDS-Unified Parkinson's Disease Rating Scale | 6 weeks
  This is an extensive scale employed for the clinical evaluation of severity of PD. It consists of four sections including non-motor findings, motor problems, motor findings, and treatment complications. Fourteen motor findings (0 - no finding, or normal, 4- severe finding) in the second section of the scale and comprising the motor problems part.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yakşi, MD, Principal Investigator — Abant İzzet Baysal University Medical Faculty
Locations (1):
- Elif Yakşi, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No